CLINICAL TRIAL: NCT01356446
Title: Impact of the Surgical Checklist on 30-day and 90-day Mortality in Elective Non-cardiac Surgery
Brief Title: Checklist Application and Mortality
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital of Bolzano (Other)
Responsible Party: Principal Investigator, Matthias Bock, Impact of the Surgical Checklist on 30-day and 90-day Mortality in Elective Non-cardiac Surgery, Regional Hospital of Bolzano
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: check4outcome3
Record Dates: First submitted 2011-05-16; First posted 2011-05-19 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Mortality; Outcome
Keywords: safety; team; team performance; surgery; outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- before surgical checklist (No Intervention)
- after implementation surgical checklist (Active Comparator)
  Interventions: Procedure: implementation surgical checklist

INTERVENTIONS:
Procedure: implementation surgical checklist — a checklist according to the suggestions raised by the WHO is implemented
  Arms: after implementation surgical checklist

SUMMARY:
The study investigates the impact of the implementation of a surgical checklist on the mortality 30 days and 90 days after surgery. Patients scheduled for elective surgical procedures (excluding cardiac surgery) lasting at least 15 minutes are eligible. Surgery is performed in a single tertiary care center. The study is an open trial before and after intervention (implementation of the checklist "safe surgery saves lifes").

ELIGIBILITY:
Inclusion Criteria:

* elective surgery in general or regional anesthesia lasting > 15 min

Exclusion Criteria:

* urgent / emergent surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Change in over all mortality | within 90 days

SECONDARY OUTCOMES:
change in over all mortality | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Bock, MD, Principal Investigator — Central Hospital Bolzano, Italy
Locations (1):
- Bolzano Central Hospital, Bolzano, Italy